CLINICAL TRIAL: NCT01212445
Title: A Randomized, Open-Label, Dose-Finding Trial of Polyethylene Glycol 3350 Laxative Plus Electrolytes for the Treatment of Constipation
Brief Title: Dose-Finding Trial of Polyethylene Glycol 3350 Laxative Plus Electrolytes for the Treatment of Constipation (Protocol P07515)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18129; 2010-021367-32 (EudraCT Number)
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Electrolytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG + E, 13.125 g (Experimental): Single sachet of PEG+E (13.125 g) dissolved in 125 mL of non-carbonated water ingested orally with entire volume taken at one time
  Interventions: Drug: PEG 3350 laxative plus electrolytes (PEG + E)/Macrogol (Movicol®, BAY81-8430)
- PEG + E, 26.25 g (Experimental): Two sachets of PEG+E (26.25 g) dissolved in 250 mL of non-carbonated water ingested orally with entire volume taken at one time
  Interventions: Drug: PEG 3350 laxative plus electrolytes (PEG + E)/Macrogol (Movicol®, BAY81-8430)
- PEG + E, 39.375 g (Experimental): Three sachets of PEG+E (39.375 g) dissolved in 375 mL of non-carbonated water ingested orally with entire volume taken at one time
  Interventions: Drug: PEG 3350 laxative plus electrolytes (PEG + E)/Macrogol (Movicol®, BAY81-8430)

INTERVENTIONS:
Drug: PEG 3350 laxative plus electrolytes (PEG + E)/Macrogol (Movicol®, BAY81-8430) — 13.125 g of PEG 3350 powder with approximately 0.6 g of electrolytes

SUMMARY:
The primary objective of the study was to evaluate the proportion of subjects with a bowel movement (BM) without straining or without hard and/or lumpy stool within the first 24 h of treatment for subjects taking 1 of 3 single doses of Polyethylene Glycol (PEG) plus Electrolytes (PEG+E) (13.125 g, 26.25 g, 39.375 g). The doses specified relate to the doses of PEG. Secondary objectives were measured by analysis of a subject diary and self-reported BM data. The secondary objectives included comparisons of PEG+E doses at 24 h for: BM control; relief of gas; relief of bloating; and relief of abdominal discomfort/cramping.

In addition, the proportion of subjects with a BM (without straining and without hard and/or lumpy stool) within the first 24 h of treatment for subjects taking different doses of PEG+E was evaluated for the time to first BM.

ELIGIBILITY:
Inclusion Criteria:

* A willingness to participate in the study and comply with its procedures
* Must be ambulatory
* Male or female subjects aged 18 years or older who met two or more of the following modified Rome III-based criteria for constipation: (a) straining during at least 25% of defecations; (b) lumpy or hard stools in at least 25% of defecations; (c) sensation of incomplete evacuation for at least 25% of defecation; (d) sensation of anorectal obstruction/blockage for at least 25% of defecations; (e) manual maneuvers to facilitate at least 25% of defecations (eg, digital evacuation, support of the pelvic floor), and (f) fewer than 3 defecations per week
* Criteria fulfilled for the last 3 months with symptom onset at least 6 mo prior to diagnosis
* Had a self reported or documented history of chronic constipation
* Agreed not to use laxatives other than the study treatment from baseline/informed consent to end-of-study
* Agreed to maintain a similar diet from the week before Visit 3 to the end-of-study were to be enrolled
* Additionally required not to use any treatment known to cause constipation during the study (for subjects enrolled after Amendment 1)
* If a female subject, either surgically sterile, 2 years postmenopausal, or using an acceptable method of contraception. Abstinence was not an acceptable method of contraception. Females of childbearing potential had to have a urine pregnancy test (human chorionic gonadotropin [HCG]) that was negative at Visit 3
* Be able to read and write in the diaries in English

Exclusion Criteria:

* Had loose stools without the use of laxatives
* Recurrent abdominal pain
* Known or suspected bowel perforation, obstruction, or fecal impaction; or had gastric retention, inflammatory bowel disease, bowel resection, or colostomy
* Celiac disease or known gluten sensitivity
* Known renal or hepatic insufficiency
* Recent history of alcohol abuse or drug abuse
* History of psychiatric disorders
* History of significant ongoing medical problems or scheduled for surgical procedures
* Subjects who, in the opinion of the Investigator, should not have been included in the study for any reason, including inability to follow study procedures
* Participated in an investigational clinical, surgical, drug or device study within the past 30 days
* Pregnant or lactating
* Allergic to PEG or PEG+E
* Employed by or have immediate family members employed by a company that manufactures laxative products
* Participant or family member of the Investigator or site staff directly involved with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cork, Ireland

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG + E 13.125 g: Participants received Polyethylene Glycol plus Electrolytes (PEG+E) as a single sachet of PEG+E (13.125 g) dissolved in 125 mL of non-carbonated water ingested orally with entire volume taken at one time on the day of open-label treatment.
- PEG + E 26.25 g: Participants received Polyethylene Glycol plus Electrolytes (PEG+E) as two sachets of PEG+E (26.25 g) dissolved in 250 mL of non-carbonated water ingested orally with entire volume taken at one time on the day of open-label treatment.
- PEG + E 39.375 g: Participants received Polyethylene Glycol plus Electrolytes (PEG+E) as three sachets of PEG+E (39.375 g) dissolved in 375 mL of non-carbonated water ingested orally with entire volume taken at one time on the day of open-label treatment.
Period: Overall Study
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Started | 52 | 51 | 51
Completed | 52 | 51 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g | Total
Number analyzed (Participants) | 52 | 51 | 51 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (16.31) | 50.4 (14.27) | 43.3 (13.8) | 46.5 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 41 | 133
  Male | 4 | 7 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Bowel Movement (BM) Within 24 Hours of PEG + E Administration
Description: A successful BM was defined as a BM with no straining or hard/lumpy stools.
Time Frame: From time of study drug treatment up to 24 hours
Population: Intent-to-Treat (ITT) Population: defined as all participants randomized regardless of whether they had taken study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants | 19.2 | 31.4 | 19.2
Statistical Analysis 1: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; The treatment success rate was defined as the number of participants in a treatment group with treatment successes (BM with no straining or hard/lumpy stools) divided by the total number of participants in the treatment group. Treatment success rate was calculated for each dose group along with 95% confidence intervals (CI) based on exact binomial statistics. Treatment success rates were compared between each pair of treatments using an exact 2-sided test (Fisher's); Test type: Superiority or Other; p = 0.1790, Fisher Exact; Treatment Success Rate = 0.192, 95% CI 2-sided [0.096 to 0.325]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; The treatment success rate was calculated as the number of participants in a treatment group with treatment successes (BM with no straining or hard/lumpy stools) divided by the total number of participants in the treatment group. Treatment success rate was calculated for each dose group along with 95% confidence intervals (CI) based on exact binomial statistics. Treatment success rates were compared between each pair of treatments using an exact 2-sided test (Fisher's); Test type: Superiority or Other; p = 1.0000, Fisher Exact; Treatment Success Rate = 0.314, 95% CI 2-sided [0.191 to 0.459]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2558, Fisher Exact; Treatment Success Rate = 0.196, 95% CI 2-sided [0.098 to 0.331]
Statistical Analysis 4: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; Logistic regression analysis was performed with treatment success as the dichotomous dependent variable and dose (13.125g, 26.25g, or 39.375 g) as the independent variable. The main effects for the model were tested for significance at the 5% level. The odds of response for the 26.25 g dose level versus the 13.125 g dose level were presented together with the associated 95% confidence interval. There were no multiplicity adjustments; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.920, 95% CI 2-sided [0.774 to 4.763]
Statistical Analysis 5: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; Logistic regression analysis was performed with treatment success as the dichotomous dependent variable and dose (13.125g, 26.25g, or 39.375 g) as the independent variable. The main effects for the model were tested for significance at the 5% level. The odds of response for the 39.375 g dose level versus the 13.125 g dose level were presented together with the associated 95% confidence intervals. There were no multiplicity adjustments; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.024, 95% CI 2-sided [0.386 to 2.720]

2. Secondary Outcome: Number of Participants With Time To First Successful BM In 0 Days Through 0.5 Days, >0.5 Days Through 1.0 Days, or >1.0 Days Through 1.5 Days After PEG+E Administration
Description: Time to first successful bowel movement was defined as the duration (in days) from the time of first study dose of study treatment until first successful BM (defined as BM without straining and without hard and/or lumpy stool).
Time Frame: From time of study drug administration up to 3 Days
Population: Participants in the ITT Population (defined as all participants who were randomized regardless of whether they had taken study treatment) who had a successful bowel movement (no straining or hard/lumpy stools). Participants who reported no successful BMs were censored.
Measure: Number; unit: participants
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 11 | 16 | 12
participants
  Successful BM in 0 days through 0.5 days | 4 | 8 | 6
  Successful BM in >0.5 days through 1.0 days | 6 | 8 | 4
  Successful BM in >1.0 days through 1.5 days | 1 | 0 | 2

3. Secondary Outcome: Percentage of Participants With Successful BM Within 12 Hours of PEG+E Administration
Description: A successful BM was defined as a BM with no straining or hard/lumpy stools.
Time Frame: From time of study drug treatment up to 12 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 52 | 51 | 51
percentage of participants | 7.7 | 15.7 | 11.8
Statistical Analysis 1: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2350, Fisher Exact; Treatment Success Rate = 0.077, 95% CI 2-sided [0.021 to 0.185]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5256, Fisher Exact; Treatment Success Rate = 0.157, 95% CI 2-sided [0.070 to 0.286]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7746, Fisher Exact; Treatment Success Rate = 0.118, 95% CI 2-sided [0.044 to 0.239]
Statistical Analysis 4: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; Logistic regression analysis was performed with treatment success as the dichotomous dependent variable and dose (13.125g, 26.25g, or 39.375 g) as the independent variable. The main effects for the model were tested for significance at the 5% level. The odds of response for the 26.25 g dose level versus the 13.125 g dose level were presented together with the associated 95% confidence intervals. There were no multiplicity adjustments; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 2.233, 95% CI 2-sided [0.628 to 7.940]
Statistical Analysis 5: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.600, 95% CI 2-sided [0.424 to 6.043]

4. Secondary Outcome: Mean Visual Analog Scale (VAS) Rating for BM Control
Description: The VAS is a psychometric response scale which measures responses along a continuum of values. The BM control VAS uses a 100 mm horizontal line with the two ends representing the opposite, extreme limits of the participant's experience of BM control. Participants marked where they felt they resided between the two ends with a vertical line. The distance from the left end of the VAS (0 mm) to the participant's mark was measured and recorded in mm. BM Control ratings ranged on a continuous scale from 0 to 100 mm, where 0 mm=Calm, not urgent and 100 mm= Not able to hold BM, very urgent.
  Participants completed a VAS after every BM or attempted BM. The VAS ratings recorded in the diaries for each BM were averaged (with range) to yield a single score for each participant. Participant scores were then averaged by treatment group
Time Frame: From time of study drug treatment up to 24 hours
Population: Participants in the ITT Population (defined as all participants who were randomized regardless of whether they had taken study treatment) who had data available.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 36 | 37 | 39
mm | 31.1 (27.27) | 23.5 (23.76) | 29.4 (23.59)
Statistical Analysis 1: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; Test type: Superiority or Other; p = 0.1876, ANCOVA; Mean Difference (Final Values) = 7.752, 95% CI 2-sided [-3.834 to 19.338]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.7680, ANCOVA; Mean Difference (Final Values) = 1.706, 95% CI 2-sided [-9.729 to 13.141]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.2941, ANCOVA; Mean Difference (Final Values) = -6.046, 95% CI 2-sided [-17.412 to 5.320]

5. Secondary Outcome: Mean VAS Rating for Gas
Description: The VAS is a psychometric response scale which measures responses along a continuum of values. The Gas VAS uses a 100 mm horizontal line with the two ends representing opposite, extreme limits of the participant's experience with BM-related gas. Participants marked where they felt they resided between the two ends with a vertical line. The distance from the left end of the VAS (0 mm) to the participant's mark was measured and recorded in mm. Gas ratings ranged on a continuous scale from 0 to 100 mm, where 0 mm=None and 100 mm= Severe.
  Participants completed a VAS after every BM or attempted BM. The VAS ratings recorded in the diaries for each BM were averaged (with range) to yield a single score for each participant. Participant scores were then averaged by treatment group.
Time Frame: From time of study drug treatment up to 24 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 39 | 40 | 42
mm | 23.9 (21.87) | 25.4 (27.14) | 26.0 (22.93)
Statistical Analysis 1: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; Test type: Superiority or Other; p = 0.8109, ANCOVA; Mean Difference (Final Values) = -1.302, 95% CI 2-sided [-12.059 to 9.454]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.6995, ANCOVA; Mean Difference (Final Values) = -2.075, 95% CI 2-sided [-12.693 to 8.544]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.8850, ANCOVA; Mean Difference (Final Values) = -0.772, 95% CI 2-sided [-11.329 to 9.784]

6. Secondary Outcome: Mean VAS Rating for Bloating
Description: The VAS is a psychometric response scale which measures responses along a continuum of values. The Bloating VAS uses a 100 mm horizontal line with the two ends representing opposite, extreme limits of the participant's experience with BM-related bloating. Participants marked where they felt they resided between the two ends with a vertical line. The distance from the left end of the VAS (0 mm) to the participant's mark was measured and recorded in mm. Bloating ratings ranged on a continuous scale from 0 to 100 mm, where 0 mm=None and 100 mm= Severe.
  Participants completed a VAS after every BM or attempted BM. The VAS ratings recorded in the diaries for each BM were averaged (with range) to yield a single score for each participant. Participant scores were then averaged by treatment group.
Time Frame: From time of study drug treatment up to 24 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 39 | 38 | 39
mm | 33.9 (32.39) | 21.7 (25.10) | 32.7 (29.55)
Statistical Analysis 1: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; Test type: Superiority or Other; p = 0.0486, ANCOVA; Mean Difference (Final Values) = 12.886, 95% CI 2-sided [0.078 to 25.695]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.8465, ANCOVA; Mean Difference (Final Values) = 1.245, 95% CI 2-sided [-11.471 to 13.962]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.0744, ANCOVA; Mean Difference (Final Values) = -11.641, 95% CI 2-sided [-24.449 to 1.167]

7. Secondary Outcome: Mean VAS Rating for Abdominal Discomfort/Cramping
Description: The VAS is a psychometric response scale which measures responses along a continuum of values. The Abdominal Discomfort/Cramping VAS uses a 100 mm horizontal line with the two ends representing opposite, extreme limits of the participant's experience with BM-related abdominal discomfort/cramping. Participants marked where they felt they resided between the two ends with a vertical line. The distance from the left end of the VAS (0 mm) to the participant's mark was measured and recorded in mm. Abdominal discomfort/cramping ratings ranged on a continuous scale from 0 to 100 mm, where 0 mm=None and 100 mm= Painful.
  Participants completed a VAS after every BM or attempted BM. The VAS ratings recorded in the diaries for each BM were averaged (with range) to yield a single score for each participant. Participant scores were then averaged by treatment group.
Time Frame: From time of study drug treatment up to 24 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 37 | 38 | 41
mm | 17.4 (24.91) | 14.0 (22.56) | 14.5 (16.89)
Statistical Analysis 1: Comparison: PEG + E 26.25 g; Test type: Superiority or Other; p = 0.4591, ANCOVA; Mean Difference (Final Values) = 3.690, 95% CI 2-sided [-6.153 to 13.534]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.5546, ANCOVA; Mean Difference (Final Values) = 2.887, 95% CI 2-sided [-6.765 to 12.539]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.8685, ANCOVA; Mean Difference (Final Values) = -0.803, 95% CI 2-sided [-10.397 to 8.790]

8. Secondary Outcome: Mean Participant Global Assessment of Treatment
Description: At the End of Study Visit, the study staff asked the participant to rate their global assessment of the study treatment according to the following categories: 0 = not at all effective, 1 = a little bit effective, 2 = moderately effective, 3 = quite a bit effective, 4 = extremely effective.
Time Frame: From time of study drug administration up to 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Number analyzed (Participants) | 52 | 51 | 51
units on a scale | 1.0 (1.15) | 1.3 (1.26) | 1.2 (1.20)
Statistical Analysis 1: Comparison: PEG + E 13.125 g vs PEG + E 26.25 g; Test type: Superiority or Other; p = 0.1865, ANCOVA; Mean Difference (Final Values) = -0.311, 95% CI 2-sided [-0.774 to 0.152]
Statistical Analysis 2: Comparison: PEG + E 13.125 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.5530, ANCOVA; Mean Difference (Final Values) = -0.139, 95% CI 2-sided [-0.602 to 0.323]
Statistical Analysis 3: Comparison: PEG + E 26.25 g vs PEG + E 39.375 g; Test type: Superiority or Other; p = 0.4670, ANCOVA; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [-0.293 to 0.637]

ADVERSE EVENTS:
Arm/Group | PEG + E 13.125 g | PEG + E 26.25 g | PEG + E 39.375 g
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Schering-Plough HealthCare Products, Inc. reserves all publication and presentation rights.